## **Analysis Plan**

Unique Protocol ID: EtikDnr2021-04357CUST1

Brief Title: Self-compassion Therapist-led Online Group Treatment for Adolescents With

Distress, Anxiety, and Depression (CUST)

Official Title: The Effects of a Self-compassion Therapist-led Online Group Treatment for

Adolescents With Distress, Anxiety and Depression

NCT number: 05448014 Document date: 1 July 2022

## Data calculations

To address outcomes, data will be screened for faulty values and dependent variables will be examined for normality.

Randomization exclude systematic differences between groups (CFT group (n=17) and control group (n=17, waitlist)) at baseline, so the investigators will only calculate differences in effect sizes (Hedge g and Cohens d) on baseline demographic and psychosocial variables.

Descriptive statistics will be calculated for CFT group and control group for pre- and post-intervention.

To assess whether the groups (CFT group and control group) differ on post values, the investigators will conduct three Ancovas controlling for baseline. Dependent variables: posttest of total score of Perceived Stress Scale, subscale anxiety and depression in Trauma Symptom Checklist for Children (TSCC). Independent variable: Groups (CFT group and control group). Controlling variables: pretest of total score of total score of Perceived Stress Scale, subscale anxiety and depression in Trauma Symptom Checklist for Children (TSCC).

The investigators will calculate Hedges' g scores for effect size of differences between groups. Hedges' g is similar to Cohen's d, but includes a correction factor for small samples. Nonsignificant differences with Hedges' g greater than .20 are considered meaningful and are interpreted according to convention: .20=small, .50=medium, .80=large.

Finally, several Ancovas will be conducted to examine whether differences between CFT group and control group changes in secondary outcomes were found.

The investigators will use an exploratory approach for not missing any changes and the significance level will be 0.05. This study will be underpowered, and the outcome will be used

to calculate power for a larger RCT-study. The investigators will both calculate result for intention to treat and for those who have participated more than two times.

Within-participant change will be calculated with Reliable Change Index (Blampied et al., 2016).

## Reference

Blampied, N. M., Conference, N., & Wellington. (2016). Reliable change & the reliable change index in the context of evidence-based practice: A tutorial review.